CLINICAL TRIAL: NCT02220608
Title: A Phase I Study of the Safety and Feasibility of Bortezomib in Combination With G-CSF for Stem Cell Mobilization in Patients With Multiple Myeloma
Brief Title: Phase I Study of Bortezomib With G-CSF for Stem Cell Mobilization in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201412026; 1KL2TR002346-01 (NIH)
Record Dates: First submitted 2014-08-15; First posted 2014-08-20 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; G-CSF; Bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Dose Level 1 (Bortezomib & G-CSF) (Experimental): G-CSF will be administered daily for 5 days (Days 1-5). On Day 4 at approximately 1800 hours, bortezomib will be administered. Apheresis will begin on Day 5 either 15 or 18 hours following Day 4 bortezomib dose; 20L of peripheral blood will be processed with a cumulative target collection goal of > 6.0x106 CD34+cells/kg. If the target collection goal is not met after one apheresis procedures, up to three additional days of G-CSF and apheresis may be repeated.
  Interventions: Biological: Bortezomib; Drug: G-CSF
- Arm 2: Dose Level 2 (Bortezomib & G-CSF) (Experimental): G-CSF will be administered daily for 5 days (Days 1-5). On Day 4 at approximately 1800 hours, bortezomib will be administered. Apheresis will begin on Day 5 either 15 or 18 hours following Day 4 bortezomib dose; 20L of peripheral blood will be processed with a cumulative target collection goal of > 6.0x106 CD34+cells/kg. If the target collection goal is not met after one apheresis procedures, up to three additional days of G-CSF and apheresis may be repeated.
  Interventions: Biological: Bortezomib; Drug: G-CSF

INTERVENTIONS:
Biological: Bortezomib
  Other Names: Velcade; LDP 341; MLN341; PS-341
Drug: G-CSF
  Other Names: Neupogen; filgrastim XM02; granulocyte colony-stimulating factor; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; tbo-filgrastim; tevagrastim

SUMMARY:
The purpose of this research study is to determine the highest dose of a drug called bortezomib that can be given with a drug called G-CSF before stem cell collection to help in the mobilization of stem cells.

DETAILED DESCRIPTION:
The purpose of this phase I study is to define the maximum tolerated dose of bortezomib and its mobilization effects when given with G-CSF for stem cell mobilization in multiple myeloma patients. We hypothesize that bortezomib, in addition to increasing the number of mobilized stem cells, will optimize final apheresis product by decreasing myeloma cell contamination. Therefore, all multiple myeloma patients rather than multiple myeloma patients with G-CSF mobilization failure will be the target of this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of multiple myeloma.
* Eligible for autologous transplantation.
* Received at least two cycles of any regimen as initial systemic therapy for multiple myeloma and are within 2-12 months of the first dose of initial therapy.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Platelets ≥ 50,000/mm3
  * Hemoglobin ≥ 8.0 g/dL
  * Absolute neutrophil count ≥1,000/mm3
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Total bilirubin ≤ 1.5 x IULN
  * Measured or calculated creatinine clearance ≥ 30 mL/min
* Female patients who:

  * are postmenopausal for at least 1 year before the screening visit OR
  * are surgically sterile OR
  * Women of childbearing potential and men must agree to practice 2 effective methods of contraception prior to study entry, for the duration of study participation, and for 30 days after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Previous stem cell collection or transplantation (autologous or allogeneic).
* Evidence of multiple myeloma disease progression (as defined by IMWG) any time prior to auto-HSCT.
* Diagnosis of plasma cell leukemia.
* Concurrent hematologic or non-hematologic malignancy requiring treatment (other than multiple myeloma or secondary amyloidosis).
* Radiation therapy within 3 weeks prior to enrollment.
* Grade 2 or higher peripheral neuropathy.
* Known hypersensitivity to any of the following: bortezomib, boron, mannitol.
* Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, or serious medical or psychiatric illness/social situations that would limit compliance with study requirements.
* Female patients who are pregnant and/or breastfeeding. Patient must have a negative serum pregnancy test within 14 days of study entry.
* Known HIV-positivity. These patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients with HIV-positivity when indicated.
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of the trial and throughout the duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of bortezomib when given with G-CSF | Approximately 12 months (completion of all patients on trial)
  The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first 28 days after administration of the first dose of bortezomib and before auto-HSCT. Dose escalations will proceed until the MTD has been reached.

CONTACTS AND LOCATIONS:
Overall Officials: Armin Ghobadi, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghobadi A, Holt M, Ritchey J et al. The effect of Bortezomib (B) Alone or in Combination with Other Agents for Stem Cell Mobilization in Mice. Blood (ASH Annual Meeting Abstracts), Nov 2012; 120: 583
- [Derived] Ghobadi A, Fiala MA, Rettig M, Schroeder M, Uy GL, Stockerl-Goldstein K, Westervelt P, Vij R, DiPersio JF. A Phase I Study of the Safety and Feasibility of Bortezomib in Combination With G-CSF for Stem Cell Mobilization in Patients With Multiple Myeloma. Clin Lymphoma Myeloma Leuk. 2019 Oct;19(10):e588-e593. doi: 10.1016/j.clml.2019.04.017. Epub 2019 May 2. PMID 31358485
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu